CLINICAL TRIAL: NCT05023681
Title: Efficacy and Safety of an Early Phase Single Bolus r-SAK for Acute Myocardial Infarction: a Multi-center Randomized Clinical Trial (OPTIMA-5)
Brief Title: The OPTIMA-5 Trail
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chunjian Li, Chief leader of CCU, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 014
Record Dates: First submitted 2021-08-22; First posted 2021-08-26 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction；Recombinant Staphylokinase; thrombolysis
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In this study, patients are randomly assigned 1:1 to the r-SAK treatment group and the saline control group using a central randomization system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- r-SAK treatment group (Experimental): intravenous injection of single bolus 5 mg r-SAK in 3min
  Interventions: Drug: Recombinant Staphylokinase
- saline control group (Placebo Comparator): intravenous injection of 10ml saline in 3min,r-SAK and saline are the same in appearance
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Recombinant Staphylokinase — Intravenous injection of r-SAK is administered within 10 minutes after diagnosis of acute ST-segment elevation myocardial infarction
  Other Names: r-SAK single intravenous injection for early treatment of acute myocardial infarction
  Arms: r-SAK treatment group
Drug: normal saline — Intravenous injection of placebo(normal saline ) is administered within 10 minutes after diagnosis of acute ST-segment elevation myocardial infarction
  Other Names: normal saline intravenous injection for early treatment of acute myocardial infarction
  Arms: saline control group

SUMMARY:
This study was a prospective, multicenter, randomized, controlled, excellence clinical trial. Subjects meeting the inclusion/exclusion criteria were randomly assigned 1:1 to r-SAK group or the control group (normal saline). Emergency coronary angiography was performed and cardiac magnetic resonance imaging was performed 5 days after surgery, followed up to 30 days.

At present, there is still a lack of clinical evidence on whether thrombolytic therapy is performed for acute ST-segment elevation myocardial infarction <2 hours after the first medical contact and prime PCI. Compared to prime PCI, early thrombolytic therapy can undoubtedly shorten the implementation time of reperfusion strategy to the maximum. For highly effective thrombolytic drugs, it should also shorten the reperfusion time, reduce thrombotic load, possibly reduce the area of myocardial infarction and improve the prognosis of patients. In this study, normal saline was used as the control. To observe the efficacy of thrombolytic therapy with single intravenous infusion of recombinant glucokinase (r-SAK) at the first time in acute ST-segment elevation myocardial infarction. And the effect of r-SAK on improving myocardial tissue level perfusion, reducing myocardial infarction size, improving cardiac function and clinical prognosis in STEMI patients.

DETAILED DESCRIPTION:
Acute myocardial infarction (AMI) is one of the leading causes of death all over the world. Even if patients with AMI survive the acute period without death, some ones would inevitably develop into chronic heart failure due to myocardial ischemia caused by segmental ventricular wall dyskinesia, myocardial remodeling, etc., which would seriously affect the prognosis of these patients. Early intensive treatment is the decisive factor to reduce the death of patients with AMI. However, the primary hospitals where patients firstly visit do not have the ability of Primary Percutaneous Transluminal Coronary Intervention (PCI) the guidelines recommend. They have to transport patients to a center that has the conditions for emergency interventional treatment. But this transportation will delay a lot of time, resulting in the extension of MI area. More importantly, the thrombus load in coronary arteries would increase with time, and the implantation of stents in vessels with a large thrombus load will often lead to slow flow or no flow, which is a relative contraindication for interventional therapy.

At present, the guidelines recommend loading dose antiplatelet therapy and transport to the superior hospital for prime PCI within 2 hours if the first hospital for acute myocardial infarction does not have the conditions for emergency interventional therapy. Current guidelines recommend that thrombolytic therapy should be performed first and then transported when delivery is expected to be >2 hours to a hospital where PCI can be performed. And thrombolytic therapy is not recommended for patients who can perform PCI within <2 hours. There is a lack of clinical evidence for thrombolysis within 2 hours of first medical contact to Primary PCI. Compared with Primary PCI, early thrombolytic therapy can undoubtedly shorten the implementation time of reperfusion strategy to the maximum. For highly effective thrombolytic drugs, reperfusion time should be shortened, thrombus load should be reduced, and the size of myocardial infarction may be reduced and the prognosis of patients improved. There is a lack of clinical evidence for this. China is a developing country, whose grassroots and rural health resources are still poor. Early thrombolysis treatment plus subsequent reperfusion of interventional therapy not only conform to the Chinese characteristic, but also accord with the international research and the development direction in this field, which is worth further study.

Staphylokinase (SAK) is produced by Staphylococcus aureus and it is a protein containing 136 amino acid residues. Its ability for dissolving blood clots was first discovered in 1948. Studies have shown that SAK is not directly convert plasminogen (PLG) into plasminogen (PLi), but first combines with PLG in a 1:1 ratio to form a complex. The complex can lead to the exposure of PLG active site, from single chain to double chain PLi, resulting to form an active SAK-PLI complex, which subsequently activates PLG molecules. Then PLG transforms into PLi and further dissolve the thrombus.

Recombinant SAK (r-SAK) was developed in 1990 by Shanghai Institute of Plant and Biological Physiology. It is a gene recombinant drug prepared by molecular cloning of SAK gene in Escherichia coli. Its biological characteristics are very similar to natural SAK, and r-SAK is a highly fibrin-specific fibrinolysis agent. R-SAK is considered to be one of the most promising thrombolytic drugs due to its high thrombolysis activity (especially in platelet-rich arterial thrombosis), inactivation of system fibrinolysis, and few side effects. Clinical studies have shown that the efficacy of r-SAK in the treatment of AMI is better than urokinase, comparable to RT-PA, and it does not increase serious bleeding complications such as intracranial hemorrhage.

In terms of pharmacokinetics, r-SAK has a fast distribution and a long action time in human body. Half-lives of distribution term is 13.30±2.06min and elimination term is 67.94±21.39min when intravenous injection 10 mg r-SAK in 30min. A single bolus of r-SAK as early as possible during the first medical contact (such as prehospital care or primary hospitals or medical centers with conditional PCI) can maximize the time window for reperfusion therapy. R-SAK, a highly effective thrombolytic drug, may shorten the reperfusion time, reduce the size of myocardial infarction and improve the prognosis of the AMI patients.

The aim of this study was to investigate the efficacy of single bolus of r-SAK for thrombolytic therapy at the first contact with the patients who are diagnosed acute ST-segment elevation myocardial infarction. It is hypothesized that this therapy can open the culprit artery very early and effectively, reduce thrombus load, reduce slow flow or no flow caused by subsequent PCI, and improve myocardial tissue perfusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18, ≦75 years old, weight ≥45kg, gender is not limited.
2. Diagnosis of acute ST-segment elevation myocardial infarction (both of the following) (A) Ischemic chest pain lasting more than 30 minutes; (B) Ecg indicates ST-segment elevation ≥ 0.1mV in 2 or more limb leads, or ST-segment elevation ≥ 0.2mV in 2 or more adjacent chest leads;
3. Time from onset of persistent ischemic chest pain to randomization ≤12 hours;
4. Coronary angiography and/or PCI are expected to be performed within 2 hours of r-SAK thrombolysis.

Exclusion Criteria:

1. Non-ST-segment elevation myocardial infarction;
2. STEMI with cardiogenic shock;
3. active bleeding or bleeding tendency, including Ⅲ, Ⅳ period history of retinopathy, retinal hemorrhage, gastrointestinal tract and urinary tract hemorrhage (1 month), ischemic stroke happened over the past 6 months, transient ischemic attack (TIA) happened over the past 6 weeks, hemorrhagic stroke in the past, unexplained platelet count < 100 x 109 / L or Hemoglobin <100g/L;
4. Having a history of central nervous system trauma or known intracranial aneurysm;
5. Recent (within 1 month) severe trauma, surgery or head injury;
6. Suspected aortic dissection, infective endocarditis;
7. Recent history of puncture which difficult hemostasis by compression (visceral biopsy, compartment puncture);
8. Long-term use and/or current use of anticoagulant drugs;
9. Hypertension not well controlled ≥180/110mmHg;
10. Having severe hepatic and renal impairment (ALT, AST, γ-GT > 2.5 times the upper limit of normal value; Cr > 1.5 times upper normal);
11. Known allergies to r-SAK;
12. Pregnant, breastfeeding or planned pregnancy women and male patients with family planning;
13. Patients who have participated in other clinical trials in the past 3 months;
14. Having a history of myocardial infarction or CABG;
15. Having taken antiplatelet drugs after pain onset, such as clopidogrel, prasugrel, cilostazol etc;
16. Other reasons that patients considered unsuitable for inclusion by researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
the percentage of TIMI flow grade 2 and 3 or grade 3 after 60 minutes of the thrombolytic therapy | 60 minutes
  The primary endpoint
the incidence of major bleeding defined as Bleeding Academic Research Consortium (BARC) ≥3 bleeding | 30 days
  The main safety endpoint

SECONDARY OUTCOMES:
The percentage of TIMI flow grade 3 after PCI | 60 minutes
  The percentage of TIMI flow grade 3 after PCI
Clinical net benefits of MACE and major bleeding events during hospitalization | 1 week
  Clinical net benefit of MACE and major bleeding events during hospitalization
MACCEs, defined as composite of all-cause death, myocardial infarction, unplanned revascularization, ischemic stroke and cardiogenic re-hospitalization recorded during 30-day follow-up | 30 days
  MACCEs, defined as composite of all-cause death, myocardial infarction, unplanned revascularization, ischemic stroke and cardiogenic re-hospitalization recorded during 30-day follow-up
Infarct size, Microvascular obstruction, cardiac function (EF) and Intramuscular hemorrhageH detected by MRI 5 days after AMI | 5 days
  Infarct size, Microvascular obstruction, cardiac function (EF) and Intramuscular hemorrhage detected by MRI 5 days after AMI
Major bleeding (BARC ≥3) and minor bleeding (BARC ≤2) events during 30-day follow-up | 30 days
  Major bleeding (BARC ≥3) and minor bleeding (BARC ≤2) events during 30-day follow-up
The occurrence of slow or no reflow during CAG or PCI | 60 minutes
  The occurrence of slow or no reflow during CAG or PCI
Corrected TIMI Frame Count (CTFC) and TIMI Myocardial Perfusion Frame Count (TMPFC) after PCI | 60 minutes
  Corrected TIMI Frame Count (CTFC) and TIMI Myocardial Perfusion Frame Count (TMPFC) after PCI
Malignant arrhythmia after thrombolysis and during hospitalization | 1 week
  Malignant arrhythmia after thrombolysis and during hospitalization

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Changzhou Second People's Hospital, Changzhou
  - The second Affiliated Hospital of Dalian Medical University, Dalian
  - The Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou
  - Huai 'an Second People's Hospital affiliated to Nanjing Medical University, Huai'an
  - Lianyungang First People's Hospital, Lianyungang
  - Renji Hospital affiliated to Shanghai Jiaotong University, Shanghai
  - Taizhou People's Hospital, Taizhou
  - Affiliated Hospital of Jiangnan University, Wuxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Correction to: Heart Disease and Stroke Statistics-2018 Update: A Report From the American Heart Association. Circulation. 2018 Mar 20;137(12):e493. doi: 10.1161/CIR.0000000000000573. No abstract available. PMID 29555722
- [Result] Heusch G, Libby P, Gersh B, Yellon D, Bohm M, Lopaschuk G, Opie L. Cardiovascular remodelling in coronary artery disease and heart failure. Lancet. 2014 May 31;383(9932):1933-43. doi: 10.1016/S0140-6736(14)60107-0. Epub 2014 May 13. PMID 24831770
- [Result] Agnoletti G, Cargnoni A, Agnoletti L, Di Marcello M, Balzarini P, Pasini E, Gitti G, Martina P, Ardesi R, Ferrari R. Experimental ischemic cardiomyopathy: insights into remodeling, physiological adaptation, and humoral response. Ann Clin Lab Sci. 2006 Summer;36(3):333-40. PMID 16951276
- [Result] Townsend N, Wilson L, Bhatnagar P, Wickramasinghe K, Rayner M, Nichols M. Cardiovascular disease in Europe: epidemiological update 2016. Eur Heart J. 2016 Nov 7;37(42):3232-3245. doi: 10.1093/eurheartj/ehw334. Epub 2016 Aug 14. No abstract available. PMID 27523477
- [Result] Collen D, Lijnen HR. Thrombolytic agents. Thromb Haemost. 2005 Apr;93(4):627-30. doi: 10.1160/TH04-11-0724. PMID 15841305
- [Result] Pulicherla KK, Kumar A, Gadupudi GS, Kotra SR, Rao KR. In vitro characterization of a multifunctional staphylokinase variant with reduced reocclusion, produced from salt inducible E. coli GJ1158. Biomed Res Int. 2013;2013:297305. doi: 10.1155/2013/297305. Epub 2013 Aug 13. PMID 23998121
- [Result] Ueshima S, Matsuo O. Development of new fibrinolytic agents. Curr Pharm Des. 2006;12(7):849-57. doi: 10.2174/138161206776056065. PMID 16515501
- [Result] Yamamoto J, Kawano M, Hashimoto M, Sasaki Y, Yamashita T, Taka T, Watanabe S, Giddings JC. Adjuvant effect of antibodies against von Willebrand Factor, fibrinogen, and fibronectin on staphylokinase-induced thrombolysis as measured using mural thrombi formed in rat mesenteric venules. Thromb Res. 2000 Mar 1;97(5):327-33. doi: 10.1016/s0049-3848(99)00184-x. PMID 10709908
- [Result] Szemraj J, Stankiewicz A, Rozmyslowicz-Szerminska W, Mogielnicki A, Gromotowicz A, Buczko W, Oszajca K, Bartkowiak J, Chabielska E. A new recombinant thrombolytic and antithrombotic agent with higher fibrin affinity - a staphylokinase variant. An in-vivo study. Thromb Haemost. 2007 Jun;97(6):1037-45. doi: 10.1160/th06-10-0562. PMID 17549308
- [Result] Vakili B, Nezafat N, Negahdaripour M, Yari M, Zare B, Ghasemi Y. Staphylokinase Enzyme: An Overview of Structure, Function and Engineered Forms. Curr Pharm Biotechnol. 2017;18(13):1026-1037. doi: 10.2174/1389201019666180209121323. PMID 29424308
- [Result] Li CJ, Huang J, Yang ZJ, Cao KJ. Thrombolytic efficacy of native recombinant staphylokinase on femoral artery thrombus of rabbits. Acta Pharmacol Sin. 2007 Jan;28(1):58-65. doi: 10.1111/j.1745-7254.2007.00455.x. PMID 17184583
- [Result] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Result] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). Glob Heart. 2018 Dec;13(4):305-338. doi: 10.1016/j.gheart.2018.08.004. Epub 2018 Aug 25. No abstract available. PMID 30154043
- [Result] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Result] Halvorsen S, Storey RF, Rocca B, Sibbing D, Ten Berg J, Grove EL, Weiss TW, Collet JP, Andreotti F, Gulba DC, Lip GYH, Husted S, Vilahur G, Morais J, Verheugt FWA, Lanas A, Al-Shahi Salman R, Steg PG, Huber K; ESC Working Group on Thrombosis. Management of antithrombotic therapy after bleeding in patients with coronary artery disease and/or atrial fibrillation: expert consensus paper of the European Society of Cardiology Working Group on Thrombosis. Eur Heart J. 2017 May 14;38(19):1455-1462. doi: 10.1093/eurheartj/ehw454. No abstract available. PMID 27789570
- [Derived] Chen P, Eikelboom JW, Tan C, Zhang W, Xu Y, Bai J, Wang J, Wang T, Gong X, Liu K, Chen X, Wang X, Zhu L, Zhao X, Yang N, Jiang J, Pu J, Zhao B, Chen Z, Li B, Wang G, Lu C, Ying L, Jiang M, Zhu X, Ma J, Dong Z, Li C, Zong J, Zhang F, Zhu J, Huang J, Kong X, Yu H, Li C; OPTIMA-5 Investigators. Single Bolus r-SAK Before Primary PCI for ST-Segment-Elevation Myocardial Infarction. Circ Cardiovasc Interv. 2024 Feb;17(2):e013455. doi: 10.1161/CIRCINTERVENTIONS.123.013455. Epub 2024 Jan 23. PMID 38258563
- See also: Article Published in Chinese — http://en.cnki.com.cn/Article_en/CJFDTOTAL-NJYK200002004.htm